CLINICAL TRIAL: NCT02460913
Title: Acupuncture Versus Intravenous Morphine in the Management of Acute Pain in the Emergency Department. An Efficacy and Safety Study
Brief Title: Acupuncture Versus Intravenous Morphine in the Management of Acute Pain in the Emergency Department
Acronym: AcuMAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/02
Record Dates: First submitted 2015-05-25; First posted 2015-06-03 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Acute Pain
Keywords: acupuncture; morphine; acute pain
MeSH Terms: conditions — Acute Pain | interventions — Acupuncture Therapy; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): patients received a 20 to 30 minutes session of acupuncture
  Interventions: Procedure: Acupuncture
- IV Morphine (Active Comparator): patients received an intravenous titration of morphine every 5 minutes.
  Interventions: Drug: Morphine titration

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture session of 20 to 30 minutes. Treatment protocols were determined through review of major clinical manuals and textbooks, literature review, and a panel of specialist acupuncturists from Chinese medicine backgrounds.
  Arms: Acupuncture
Drug: Morphine titration — Patients in this group received IV titrated morphine. Morphine was prepared onsite and diluted in a manner to obtain a dose of 1mg in each ml of normal saline. The initial dose was 0.1 mg per kg and a titration dose of 0.05 mg per Kg was repeated every 5 minutes until reaching objective. The maximum allowed dose was 1.5 mg/kg.
  Other Names: Morphine
  Arms: IV Morphine

SUMMARY:
Inadequate pain management is a common problem encountered in ED settings. Pain relief medications use is often limited by their side effects. Evidence suggests that non pharmacologic pain relief techniques such as acupuncture can play a central role to treat pain in acute conditions, but their application is still scarce.

DETAILED DESCRIPTION:
Pain is a common cause of emergency department visits and its control remains a challenge and health priority worldwide. Many techniques were developed to control pain and to ensure patients comfort but their application is still difficult especially in emergency department (ED) settings, due to the variety of treated conditions, the non-availability of qualified practitioners and the patient's specificity. Pharmacologic methods in particular IV opioids are the most used and with regard to their rapid action with high efficacy. But the use of these drugs can be limited by their side effects. Non-pharmacologic pain relief techniques such as acupuncture have been proposed. During the second half of the twentieth century, acupuncture was established in Europe and in the last two decades, it has spread around the world. In Tunisia, acupuncture was introduced into the health system in the 90s, particularly to treat pain.

The World Health Organization (WHO) has recognized acupuncture as safe and sound therapy. A preliminary list of acupuncture indications has been reported including 43 diseases. However, the introduction of acupuncture in the treatment of pain in ED is more recent or even anecdotal. In the treatment of chronic pain, it was shown that acupuncture is comparable to morphine and that its better safety profile makes it the method of choice in some clinical conditions.

In a recent systematic review, it has been concluded that there is insufficient evidence for the use of acupuncture in the ED settings due to the paucity of randomized controlled trials and the suboptimal methodological qualities of related studies.

The aim of our study was to evaluate the efficacy and safety of acupuncture compared with morphine for the management of acute pain in ED.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset pain < 72 hours of the ED presentation
* Pain intensity ≥ 40 of the VAS or NRS (ranging from 0 for no pain to 100 for maximum imaginable pain)
* Acute musculoskeletal pain with no evidence of fracture or dislocation, including ankle and knee sprains without signs of severity (ligament rupture, laxity), shoulder and elbow tendinitis, upper and lower limb mechanical pains and lower back pain with no evidence of neurological deficit.
* Acute abdominal pain with no urging surgical intervention including renal colic and dysmenorrhea.
* Acute headache that meets the criteria of primary headache, as described by the international headache society.

Exclusion Criteria:

* Temperature > 37.7°c
* Violent mechanism of trauma
* Patients under anticoagulant drugs or with coagulation abnormalities
* Skin affections (infections, hematoma, dermatosis) that would impair the use of certain acupuncture points
* Patients that were judged enable to participate in the study at the discretion of the treating physician.
* Refusal, inability to consent.
* Inability to assess the degree of pain using the VAS or NRS
* Patients who had received analgesics in the 6 hours prior to the enrollment
* An initial pain score ≤ 40 on the VAS or NRS
* Patients who had presented to the ED in the last 24 hours with the same motif
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
change of pain severity from baseline | 10, 20, 30, 45, 60 minutes
  Change of pain score was assessed at 10, 20, 30, 45 and 60 minutes time points from the starting of the protocol.
  Pain severity was measured using the visual analogic scale (VAS) going from 10 (maximum imaginable pain) to 0 (no pain). if the VAS was not applicable to certain patients, a verbal numeric rating scale (NRS) was used instead.
  Success of treatment was defined by a drop in the pain intensity under 30.

SECONDARY OUTCOMES:
resolution time | 10, 20, 30, 45, 60 minutes
  This interval was defined by the time (in minutes) elapsed between the start of the protocol (T0) and the decrease of the pain score of at least 50% of its initial value.
adverse events | 10, 20, 30, 45, 60 minutes and until ED discharge
  Occurrence of major side effects implicates the immediate ending of the protocol, more particularly:
  * Allergic manifestations such as rush and generalized edema
  * severe hypotension defined by a drop of the systolic blood pressure under 90 mmHg or a loss of more than 20 mmHg of the initial systolic blood pressure
  * recurrent vomiting non controlled by the standard measures
  * Altered mental status
  * Uncontrolled bleeding from the site of needle insertion
  * Respiratory distress with capillary saturation under 95% or signs of pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: nouira semir, MD, Principal Investigator — University of Monastir

REFERENCES:
- [Background] Kim KH, Lee BR, Ryu JH, Choi TY, Yang GY. The role of acupuncture in emergency department settings: a systematic review. Complement Ther Med. 2013 Feb;21(1):65-72. doi: 10.1016/j.ctim.2012.12.004. Epub 2012 Dec 29. PMID 23374207
- [Background] Cohen M, Parker S, Taylor D, Smit de V, Ben-Meir M, Cameron P, Xue C. Acupuncture as analgesia for low back pain, ankle sprain and migraine in emergency departments: study protocol for a randomized controlled trial. Trials. 2011 Nov 15;12:241. doi: 10.1186/1745-6215-12-241. PMID 22085683